CLINICAL TRIAL: NCT03023787
Title: A Randomized, Double-Blinded, Safety and Pharmacokinetic Study of Escalating Single Doses of Hepalatide in Healthy Volunteers
Brief Title: Study of Hepalatide(L47) at Phase Ib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai HEP Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: L47-Ib-01
Record Dates: First submitted 2017-01-15; First posted 2017-01-18 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Hepatitis B， Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Drug and Narcotic Control

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hepalatide (Experimental): Hepalatide 4.2mg, 6.3mg and 8.4mg
  Interventions: Drug: Hepalatide
- Placebo (Placebo Comparator): Placebo 4.2mg, 6.3mg and 8.4mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hepalatide — There are three cohorts as follows 4.2mg, 6.3mg, 8.4mg. At each dose level, healthy volunteers will be received treatment drug by abdominal subcutaneous injection once a day for seven days and will be monitored for 3 days.
  Other Names: treatment drug
  Arms: Hepalatide
Drug: Placebo — There are three cohorts as follows 4.2mg, 6.3mg, 8.4mg. At each dose level, healthy volunteers will be received control drug by abdominal subcutaneous injection once a day for seven days and will be monitored for 3 days.
  Other Names: control drug
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of Hepalatide(L47) and characterize the clinical pharmacokinetics in healthy volunteers.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, dose escalating, phase Ib trial, which will be conducted in No. 302 Hospital of China. There are three cohorts at dose of 4.2mg, 6.3mg and 8.4mg. All healthy volunteers will be randomized into Hepalatide or placebo group at 4:1 rate, all healthy volunteers will be received treatment drug by abdominal subcutaneous injection once a day for seven days and will be observed for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 45 years
* BMI Index between 19 and 25 (BMI=weight/height2)
* Normal previous history and physical exam
* No drug and alcohol abuse
* No illness in 4 weeks and no drug therapy in 2 weeks
* No blood donation or subject not sampled in 3 months
* Consistent and correct use of recommended methods of birth control for men and women
* Good compliance with study protocol
* Understand and agree to sign a consent form

Exclusion Criteria:

* Infection with HAV, HBV, HCV, HEV, HIV, EBV or CMV
* Abnormal and clinical significance test of physical examination, vital signs, blood routines, urine routines, liver and kidney functions, coagulation indicator, electrolyte, glucose, blood lipid, thyroid functions, chest X-Ray, ECG, B ultrasound of gallbladder, spleen and kidney, AFP ,and CEA
* Positive for anti-Pre-S1 antibody
* Women being pregnant or nursing, or with abnormal sex hormones, B ultrasound of ovaries/uterus proliferative diseases or breast mass
* Unable to quit smoking in trial
* Subject with little chance of enrollment (i.e. the weak)
* Subject not suitable to join the trial under other circumstances judged by investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Healthy participants with treatment-related adverse events as assessed by "guiding principle of grading standards for the adverse reactions in clinical trials of vaccine for prevention" or CTCAE v4.0 | 6 months

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 6 months
Area under the plasma concentration versus time curve (AUC) | 6 months
half-time | 6 months
apparent volume of distribution | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: zhenman wei, Principal Investigator — 302 Military Hospital
Locations (1):
- 302 Military Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No